CLINICAL TRIAL: NCT00821535
Title: An Open Label Single Dose Study To Investigate Safety And Pharmacokinetics Of Maraviroc Following A Single Oral Dose Of 300 Mg Maraviroc (Two 150 Mg Maraviroc Commercial Tablets) Under Fasting Conditions In Healthy Male Japanese Volunteers
Brief Title: Investigation Of Safety And Pharmacokinetics Following A Single Oral Dose Of 300 Mg Maraviroc In Healthy Male Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: A4001084
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: pharmacokinetics, Japanese, healthy volunteer, maraviroc
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active group (Other): maraviroc dosing group
  Interventions: Drug: maraviroc (Selzentry, Celsentri)

INTERVENTIONS:
Drug: maraviroc (Selzentry, Celsentri) — 12 subjects will receive a single dose of 300 mg maraviroc (two 150 mg maraviroc commercial tablets) under fasting conditions.
  Other Names: Selzentry, Celsentri

SUMMARY:
To confirm safety and pharmacokinetics of maraviroc following a single oral dose of 300 mg maraviroc in healthy male Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Japanese subjects between the ages of 21 and 50 years inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >45 kg.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Positive result for HIV, Hepatitis B surface antigen (HbsAg) or HCV antibody.
* Hypersensitivity/allergic reactions to any component of maraviroc, including soy lecithin.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Plasma and urine maraviroc concentrations for pharmacokinetic analysis | pre-48 hrs post dose
Adverse event monitoring | Day 0 to Day 3
Bood pressure, pulse rate | Day 0, Day 1, and Day 3
Blood and urine safety laboratory tests | Day 0 and Day 3
ECG | Day 0 and Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001084&StudyName=Investigation%20Of%20Safety%20And%20Pharmacokinetics%20Following%20A%20Single%20Oral%20Dose%20Of%20300%20Mg%20Maraviroc%20In%20Healthy%20Male%20Japanese%20Volunteers